CLINICAL TRIAL: NCT07339059
Title: Phase II Study of Sacituzumab Govitecan With Atezolizumab/Durvalumab as Maintenance Therapy for Extensive-Stage Small Cell Lung Cancer
Brief Title: SG and Immunotherapy as Maintenance Therapy for Extensive-stage Small-cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bindu R Potugari (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Bindu R Potugari, Thoracic Oncologist, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFH-C-2025-02
Record Dates: First submitted 2025-10-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer ( SCLC ); Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Keywords: atezolizumab; durvalumab; sactizumab govetican; small cell lung cancer; sclc; es-sclc; lung cancer; extensive stage
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — sacituzumab govitecan; atezolizumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SG and atezolizumab/durvalumab (Experimental): Sacituzumab govitecan 10 mg/kg via IV infusion on Day 1 and Day 8 of a 21-day cycle (ie, 2 weekly doses plus 1 week without treatment)
  AND
  Atezolizumab 1200mg via IV infusion on Day 1 of a 21-day cycle (ie, once every 3 weeks)
  OR
  Sacituzumab govitecan 10 mg/kg via IV infusion on Day 1 and Day 8 of a 21-day cycle (ie, 2 weekly doses plus 1 week without treatment)
  AND
  Durvalumab 1500mg via IV infusion on Day 1 of a 21-day cycle (ie, once every 3 weeks)
  Interventions: Drug: Sacituzumab govitecan; Drug: Atezolizumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan 10 mg/kg via IV infusion on Day 1 and Day 8 of a 21-day cycle (ie, 2 weekly doses plus 1 week without treatment)
  Other Names: Trodelvy
Drug: Atezolizumab — Atezolizumab 1200mg via IV infusion on Day 1 of a 21-day cycle (ie, once every 3 weeks)
  Other Names: Tecentriq
Drug: Durvalumab — Durvalumab 1500mg via IV infusion on Day 1 of a 21-day cycle (ie, once every 3 weeks)
  Other Names: Imfinzi

SUMMARY:
The goal of this clinical trial is to learn if the combination of sacituzumab govetican (SG) and atezolizumab/durvalumab is effective in controlling cancer tumor growth in adults with extensive stage small cell lung cancer. These drugs are FDA approved individually in different cancers. This combination is evaluated in breast cancer and showed promising combination.

The effectiveness of this treatment combination will be measured by changes in tumor size and appearance of new tumors.

Participants in the trial will:

* receive treatment SG and immunotherapy every 21 days for up to 2 years or until it is no longer works for the patient.
* CT scans at 6weeks for first 6 cycles and then every 9-12 weeks and MRI brain every 12 weeks.
* provide tissue (optional) and blood for additional testing (learn about the cancer).

DETAILED DESCRIPTION:
Small Cell Lung Cancer (SCLC) is a high-grade neuroendocrine tumor, accounting for nearly 15% of all lung cancers. It is characterized by rapid doubling time, high vascularity, apoptotic imbalance, and early widespread hematogenous metastasis. More than two-thirds of the patients present with extensive stage and only one-third of them present with limited stage confined to the chest. Prognosis continues to be poor with a 3yr relative survival rate of 13%. Despite high response rate with platinum-based chemotherapy, the median survival is limited in patients with advanced SCLC due to early recurrence. The addition of atezolizumab to platinum doublet in the extensive stage has shown only marginal improvement in both progression free survival (PFS) (5.2 months vs 4.3 months) and median overall survival (OS) (12.3 months vs 10.3 months) Similar results were observed with the addition of Durvalumab (median OS- 12.9 months vs 10.5 months). Therefore, there is a significant need to develop strategies that can sustain the response of platinum-based chemotherapy and thus prolong PFS and OS in advanced SCLC patients.

Transmembrane glycoprotein Trophoblast cell surface antigen 2 (TROP-2) is expressed at membranous and/ or cytoplasmic levels in many epithelial solid tumors including SCLC and is associated with poor prognosis. It plays an important role in carcinogenesis and tumor progression. Sacituzimab govitecan (SG) is an anti-TROP-2 antibody-drug conjugate composed of a humanized monoclonal antibody coupled with a toxic payload, SN-38, an active metabolite of irinotecan with a hydrolyzable linker. The antitumor activity/ efficacy of SG in SCLC was first noticed in first in human studies with >30% reduction of target lesions even after progression on prior topoisomerase I inhibitor. SG was evaluated in a phase I/II dose expansion/ escalation cohort to assess safety and efficacy in relapsed and refractory SCLC following 2 median prior therapies with a primary endpoint of objective response, assessed by imaging. A dose of 10mg/kg was determined to be dose-maximized efficacy and safety. Key treatment-related adverse events reported were neutropenia (57.8%) and diarrhea (56.2%). Patients with homozygous UGT1A1 allele status had an increased risk of neutropenia. Other common side effects reported were nausea/ vomiting, abdominal pain, anorexia, constipation, fatigue, anemia, and alopecia. Overall response rates of 14% (7/50) based on ITT (intention to treat) and 17% (6/36) for patients in the 10 mg/kg dose group, with a median duration of response of 5.7 months. Stable disease is noted in 42% of patients (21/50). In an open-label, multicohort Phase 2 study (TROPiCS-03), SG was evaluated in a second-line setting in patients who progressed after chemotherapy/immunotherapy in SCLC. Among 43 patients enrolled, the overall response rate was 41.9%, with a median PFS of 4.4 months (95% CI 3.81-6.11) and a median OS of 13.6 months (95% CI 6.57-14.78). All patients had treatment-related adverse events, and no AE led to treatment discontinuation.

The rationale for combining SG with immunotherapy:

Antibody-drug conjugate promotes antigen uptake and migration of dendritic cells in the tumor to tumor-draining lymph nodes, promoting T cell priming, expansion, and increased infiltration in the tumor microenvironment (TME). The infiltrating cytotoxic CD8 T cells can be stimulated with an immune checkpoint inhibitor, which effectively enhances and sustains the T cell response in the TME promoting an anti-tumor effect. SG in combination with pembrolizumab was evaluated after platinum-based chemotherapy which showed higher response rates with manageable toxicity in metastatic urothelial cancer. SG combined with atezolizumab has been evaluated in other solid tumors- breast cancer.

Given the responses in relapse and refractory SCLC with single agent SG and the potential additive effect with the combination of ADC and immunotherapy, investigators hypothesize that the addition of SG to atezolizumab/durvalumab after completion of induction platinum-based chemo-immunotherapy will improve and sustain the response rates and prolong the survival. To test the hypothesis, investigators aim to assess the clinical efficacy of the combination of SG and atezolizumab/durvalumab in a phase 2 study.

This is a prospective single-arm phase 2 study aiming to evaluate the clinical efficacy of the combination of maintenance SG and atezolizumab/ durvalumab in patients with extensive stage SCLC after completion of at least 4-6 cycles of platinum-based chemotherapy and immunotherapy. Participants with either stable disease or partial response and no evidence of disease progression as per RECIST 1.1 on restaging CT chest, abdomen, pelvis, and MRI brain will be enrolled before initiation of maintenance immunotherapy. Response and disease status for study eligibility will be based on the investigator's determination per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1), and for CNS disease by mRECIST.

Eligible participants will be consented within 4 weeks after day 1 of the last cycle of chemo-immunotherapy. Patients will receive study treatment of the combination of SG at a dose of 10mg/kg on day 1 and day 8 along with atezolizumab 1200mg on day 1 every 3 weeks or Durvalumab 1500mg on day 1 every 3 weeks for 2yr or until disease progression, unacceptable toxicity, withdrawal of consent, loss of follow-up, or death, whichever comes first. Study treatment should be initiated within 3-6 weeks of the last chemo-immunotherapy after enrollment. Treatment beyond the progression may be allowed after discussion with PI if the participant continues to derive clinical benefit in the opinion of the investigator.

Safety assessments will be conducted before day 1 of each cycle. Dose modifications will be made as necessary and can occur mid-cycle if indicated or needed. Safety follow-up should occur approximately 30 days after the end of the treatment visit or before initiation of a new antineoplastic therapy, whichever occurs first. If a participant is unable to return for safety follow-up, this will not be considered a protocol deviation. Long-term follow-up will begin after safety follow-up and will follow the radiographic imaging schedule. Radiographic imaging should continue during long-term follow-up for participants who discontinue study drug treatment for any reason other than disease progression per RECIST 1.1, withdrawal of consent for follow-up, or death. Survival will be followed until death. For those who come off treatment for disease progression (or who progress during long-term follow-up), survival status will be assessed every 12 weeks via clinic visits, by phone contact, chart review, or other acceptable methods until the participant dies, withdraws consent, or the study is terminated.

The Henry Ford Cancer Data Safety Monitoring Board (DSMB) will review periodic safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female aged 18 years or above.
* Participants must have a histologically or cytologically confirmed diagnosis of small cell lung cancer (SCLC) and extensive stage at diagnosis or locally advanced disease and unable to receive curative intent radiation.
* Participants must have received at least four cycles of platinum plus etoposide and at least 2-3 cycles of atezolizumab/ Durvalumab.
* No evidence of progression on restaging CT CAP following 4-6 cycles of Chemo/IO from the last dose of the chemotherapy cycle.
* ECOG performance status of 0-2
* Patients must not have active uncontrolled HIV, HBV, and HCV infections. Well-controlled infections on treatment will be allowed to participate in the trial.
* Patients with stable and asymptomatic brain metastasis.
* Adequate organ function - bone marrow, kidney, and liver.

Exclusion Criteria:

* Significant renal impairment requiring dialysis or hepatic impairment with end-stage liver disease.
* Participants with leptomeningeal disease.
* Participants with a recent diagnosis of heart failure and acute coronary disease within 3 months.
* Participants who are unable to receive immunotherapy with chemotherapy for induction will be excluded, or those immunotherapy was discontinued to manage immune-related adverse events
* Active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months of enrolment.
* Patients with prior exposure to anti-PD-1, anti-PD-L1, or anti-PD-L2 agents or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4) within 12 months of the study is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease Control | 12 weeks from study enrollment
  To evaluate the rate of disease control at 12 weeks for patients with extensive stage small cell lung cancer treated with Sacituzumab govitecan (SG) plus atezolizumab or durvalumab as maintenance therapy after induction treatment with chemotherapy and immunotherapy.
  Disease Control at 12 weeks is defined as a best response by RECIST 1.1 of CR, PR, non-CR, non-PR, or stable disease assessed by RECIST 1.1 and reported within 12 weeks (+/- 2 weeks) from the initiation of study therapy. Participants not known to have disease control at 12 weeks will be coded as lacking disease control.

SECONDARY OUTCOMES:
Overall Survival | Through study completion, an average of 1 year
  Overall Survival (OS): OS is defined as the duration from study registration to death due to any cause. Patients last known to be alive will be censored at the date of last contact.
Progression Free Survival | Through study completion, an average of 1 year
  Progression-free survival (PFS): PFS is defined as the duration from study registration to progression, symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free will be censored at the date of [last contact or disease assessment].
Combination therapy toxicity | Through study completion, an average of 1 year
  To measure the frequency and severity of toxicity by incidence of treatment-emergent adverse events (TEAEs) and clinical laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Cancer- Detroit, Detroit, Michigan, United States